CLINICAL TRIAL: NCT02463604
Title: Renal PRotection Against Contrast mEdium-induced nephroPathy in High Risk Patients undErgoing Coronary Angiography
Acronym: PREPARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2014-A01281-46
Record Dates: First submitted 2015-06-02; First posted 2015-06-04 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Renal Insufficiency; Contrast Medium-induced Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remote Ischemic Preconditioning (Experimental): A blood pressure cuff is placed on upper arm and inflated to 200 mmHg for 5 minutes and then deflated for 5 minutes. This cycle is repeated 3 times in total.
  The procedure has to be completed between 5 and 60 minutes prior coronary angiography.
  Interventions: Procedure: Coronary Angiography
- Control (Sham Comparator): A blood pressure cuff is placed on upper arm and inflated to 10 mmHg for 5 minutes and then deflated for 5 minutes. This cycle is repeated 3 times in total.
  The procedure has to be completed between 5 and 60 minutes prior coronary angiography.
  Interventions: Procedure: Coronary Angiography

INTERVENTIONS:
Procedure: Coronary Angiography — Coronary angiography is performed following usual site standards

SUMMARY:
This study evaluates the efficacy of remote ischemic preconditioning on preventing contrast medium-induced nephropathy in a population of high risk patients undergoing coronary angiography. Half of participants will receive a preconditioning procedure while the other half will receive a sham procedure.

DETAILED DESCRIPTION:
Contrast medium-induced nephropathy has a big impact on clinical outcomes in patients suffering from renal insufficiency who undergo percutaneous coronary interventions.

Remote ischemic preconditioning is proved to protect myocardium in patients undergoing percutaneous coronary angiography.

We will evaluate the effect of remote preconditioning on renal protection.

ELIGIBILITY:
Inclusion Criteria:

1. Patient headed to coronary angiography
2. Glomerular filtration rate :

   * ≤ 40ml/min/1,73m² (MDRD equation)
   * or ≤ 60ml/min/1,73m² (MDRD equation) with 1 additional risk factor : age > 75 years, NYHA ≥ III/IV, diabetes mellitus
3. Signed informed consent

Exclusion Criteria:

1. Preoperative assessment / dilated cardiomyopathy assessment
2. Acute ST-segment elevation myocardial infarction
3. Cardiogenic shock requiring pressor amine or systolic blood pressure <80mmHg
4. Resuscitation after cardiac arrest
5. Intra-aortic balloon pump
6. Contraindication for the repeted use of an upper-arm pressure cuff
7. Extra-renal epuration
8. No health insurance coverage
9. Legal incapacity (patients under tutorship, curatorship or judicial protection)
10. Patient enrolled in another interventional trial or being in a washout period
11. Incapacity/impossibility to undergo 12-month follow-up
12. Patient refusal

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2015-06; Primary Completion 2016-02 (Actual); Study Completion 2017-03-24 (Actual)

PRIMARY OUTCOMES:
Increase in serum creatinin level (≥25% or 0,5mg/dL) | 48h after coronary angiography
  Serum creatinin level is measured 48h after coronary angiography to assess contrast medium-induced nephropathy

SECONDARY OUTCOMES:
Serum creatinin level is measured 12 months after coronary angiography and major adverse events are collected to assess long-term effects of remote ischemic preconditioning on renal function | 12 months after coronary angiography

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Prunier, Professor, Principal Investigator — UH Angers, Cardiology
Locations (1):
- UH Angers - Cardiology ward, Angers, France